CLINICAL TRIAL: NCT01234220
Title: Multicenter Study on Use and Interpretation of Adrenal Vein Sampling
Brief Title: Adrenal Vein Sampling International Study (AVIS Study)
Acronym: AVIS
Status: Completed | Type: Observational
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, MD, FAHA, FACC, University Hospital Padova
Other Study IDs: GPR-AVIS
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Hyperaldosteronism
Keywords: Aldosterone; Primary Aldosteronism; Aldosterone Producing Adenoma (APA); Idiopathic Adrenal Hyperplasia (IHA); Adrenal Venous Sampling
MeSH Terms: conditions — Hyperaldosteronism; Adrenocortical Adenoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adrenal Venous Sampling (AVS): Patients with Primary Aldosteronism (PA) undergoing AVS to discriminate PA forms with unilateral from bilateral excess aldosterone production.

SUMMARY:
The AVIS Study is a retrospective multicenter international study that aims to answer a series of questions on the use and performance of adrenal venous catheterization (AVS) for the diagnosis of primary hyperaldosteronism subtype. A questionnaire will be circulated among the centres that are internationally recognized and have published in the field of AVS and have agreed to participate in the study.

The first aim of the AVIS study is to collect summary data on how AVS is being performed throughout the world to answer the following questions:

* How many AVS studies haw been performed yearly from 2005 to 2010 at each center?
* How many adrenal vein ruptures occurred during the AVS at each center?Has the rate of adrenal vein rupture been steady or has it changed over the 5 years?
* How many centers use bilaterally simultaneous and how many use sequential AVS catheterization?
* How many radiologists perform AVS at each center?
* How many centers use a cosyntropin stimulation during AVS?
* What is the percentage of PA patients in whom AVS is performed?
* How many centres calculate the selectivity index? What is the minimum cutoff used?
* How many centers calculate the lateralization index? What is the minimum cutoff used?
* Are the AVS studies that are not bilaterally selective used for diagnosis?
* How many centers calculate the controlateral suppression index and what is the minimum cutoff used?
* What is the cost of AVS for the National Health System or Insurance and for patients? The second aim of the study is to calculate the rate of AVS studies that are selective and show lateralization of aldosterone excess at each center by applying predefined set of criteria for defining selectivity and lateralization. Data on the final diagnosis of the PA subtype will be gathered and used as reference to assess the performance of AVS using receiver operating characteristic curves analysis and the Youden index to determine the optimal cutoffs. A worksheet will need to be completed providing information on the following: Demography; Date of AVS;Baseline blood pressure (BP) values and serum K+;Dynamic test during the AVS if any; plasma aldosterone and cortisol concentration in the infra-adrenal inferior vena cava and in the right and left adrenal vein; diagnosis of PA subtype; treatment (adrenalectomy or pharmacological therapy); post-treatment BP and serum K+ values; concordance/discordance between imaging (CT or RM) and AVS.

DETAILED DESCRIPTION:
Background. AVS is recommended by the current Endocrine Society Guideline as the gold standard for the identification of the surgically curable subtype of primary aldosteronism (PA).(Funder 2008) However, consensus on the way AVS should be performed and on the interpretation of its results still lacks, as recently pointed out. (Stewart 2010, Auchus 2010) In particular, some centers use the bilateral simultaneous technique, while others perform the sequential catheterization. Moreover, some centers perform AVS during or after using ACTH stimulation, albeit with different doses, and others do not use any stimulation.(Seccia 2009) In addition, some are utilizing the absolute values of plasma cortisol and aldosterone to determinate the lateralization (Nishikawa 2007), whereas others are relying on calculation of the selectivity index to determine the collection of adrenal vein blood, followed by calculation of the and the lateralization index only if bilaterally selective samples were obtained.(Rossi 2008) Moreover, large differences in the cutoffs for establishing selectivity and lateralization exist, which have not been clarified by recent studies that rather added further complexity to this field.(Mulatero 2010) If a consistent degree of success rate can be achieved by having only one or two radiologists performing AVS at each centre, or if more radiologists can become proficient in performing the procedure and consistently achieving adequate results, also remains to be clarified. Finally, some centers perform AVS in all patients who are plausible candidates to adrenalectomy, while other submit to AVS only a small proportion of the patients (Young WJ personal communication).

Thus, it remains unclear which is the proportion of patients with PA who are offered AVS at the different centers, and how many of those who are submitted to AVS ultimately undergo adrenalectomy.

In an era of shrinking budget the issue of cost the issue of costs of the procedure also remains a relevant one when assessing the cost-effectiveness of the diagnostic work-up of PA. A preliminary survey suggests that there are huge variations across different countries in the charges for AVS to both the patients and/or the health care and insurance system.

It is likely that one of the reasons for the lack of consensus on AVS could depend on the facts that: i) no single centre as gathered a number of AVS studies large enough to warrant solid conclusions; ii) there has been no systematic survey of the AVS data that have been generated around the world in this field

Aims of the study. Based on this background, the aims of the AVIS study are those described above.

Study design. To the first aim a questionnaire will be circulated among the centers that are internationally recognized and have published in the field of AVS and have agreed to participate in the study.

The data will be collected and handled at the maximum level of confidentiality under the requirement of the Declaration of Helsinki.

Study selection criteria. Eligible centers will be identified among those that have published in the English literature on AVS or PA (reported variously as observational cohort studies, or clinical trials): Studies will be identified through computer-assisted literature searches of databases, scanning of reference lists, hand-searching of relevant journals, correspondence with authors of relevant reports and consultation with experts in the field.

The inclusion criteria will be the consent of the leading investigator to participate in the data collection.

The only exclusion criteria will be the refusal to participate in the study. The number of adhering and non-adhering centers will be recorded and mentioned in the publications.

Data collection. Data will be collected in an anonymous way on many characteristics at baseline and at subsequent surveys during follow-up. Information on categorical variables, will be systematically re-coded to ensure comparability among studies. For each individual patient, data were sought on the following outcomes: blood pressure and antihypertensive medications at follow-up post-adrenalectomy and on dates of occurrence of cardiovascular events, including non-fatal CHD; non fatal stroke; specific cause mortality (or at least fatal CDH and fatal stroke) and other cardiovascular outcomes. Being a retrospective study, precise details of the diagnostic criteria used for the definition of incident cases will be sought from each centre (as were data on the completeness of follow-up).

Data obtained from each participating study will be checked for internal consistency and any queries that might arrive will clarified with the P.I. of each centre, before harmonization to a standard format.

The content of the data will be unchanged by this process, and computer-generated detailed summary tabulations based will be reviewed and confirmed by collaborators.

Data will be stored securely and anonymously at the coordinating centre.

Statistical analysis will be performed by use of summary statistics after appropriate transformation of the variables that show a skewed distribution as PAC and PCC by means of the SPSS for Mac (vers 18.0), GaphPad and the MedCalc softwares.

Scientific Committee. The leading investigator of each centre contributing at least 50 AVS studies will be invited to participate in the scientific committee of the AVIS study and will have full access to the locked database.

Expected results. Upon completion of the first phase of the study the investigators expect to be able to gather information on the way AVS is being performed around the world and therefore to prepare a first manuscript reporting on the number of AVS per centre, the rate of adrenal vein ruptures during the procedure, the rate of use of simultaneous/sequential AVS catheterization, the number of radiologists that perform AVS and their success rate in the procedure, the rate of use of stimulation test during the perform of AVS, the percentage of PA patients to whom AVS is offered at each center, the rate of calculation of the selectivity index, the lateralization index and the contralateral suppression index and their cutoff limits, the use of AVS studies that are not bilaterally selective for diagnosis and the costs of AVS for the National Health System or Insurance and for the patients.

Upon completion of the database with the individual data the investigators expect to be able to gather > 2000 AVS studies, in a single database. After harmonization of the data, identification of the outliers and of the underlying reasons (by interaction with the leading investigator at each center), the database will be locked. The investigators will then undertake the statistical analysis, which will entail the following variables:

* Demography (sex, age, race);
* Baseline blood pressure (BP) and heart rate (HR) values;
* Serum K+ before AVS;
* Dynamic test during the AVS if any;
* Plasma aldosterone (PAC) and cortisol concentration (PCC) in the infraadrenal inferior vena cava (IVC) and in the right (RAV) and left (LAV) adrenal vein;
* Final diagnosis (bilateral adrenocortical hyperplasia (BAH), unilateral adrenocortical hyperplasia (UAH), aldosterone-producing adenoma (APA), bilateral APA;
* Treatment (adrenalectomy or pharmacological therapy);
* Post-treatment blood pressure (BP) and heart rate (HR) values;
* Post-treatment sK+ ;
* Diagnosis concordance/discordance between imaging (CT or RM) and AVS. Data on the demography, biochemical and hemodynamic features of the patients selected for AVS in the different continents will be obtained and information on the rate of successful catheterization will be generated. The concordance rate of imaging and AVS results will also be determined and the clinical usefulness of the AVS for establishing the indication to adrenalectomy will be ascertained in the largest database available ever.

ELIGIBILITY:
Inclusion Criteria:

* consent of the leading investigator to participate to the data collection

Exclusion Criteria:

* refusal of the leading investigator to participate to the AVIS Study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with Primary Aldosteronism who underwent AVS during the last 5 years in 15 worldwide centers.
Sampling Method: Non-Probability Sample
Enrollment: 2604 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Number of adrenal vein ruptures occurring during AVS | January 1st 2005 - November 1st 2010

SECONDARY OUTCOMES:
AVS cost for the patient and the health insurance system | January 1st 2005 - November 1st 2010
  The amount in euros that the patient and the health insurance system has to pay for the AVS study will be estimated in each center.
number of selective AVS at right or left side | January 1st 2005 - November 1st 2010
  The number of selective AVS at right or left side will be calculated using different cutoff values for the selectivity index.
number of bilaterally selective AVS | January 1st 2005 - November 1st 2010
  The number of bilaterally selective AVS will be calculated using different cutoff values for the selectivity index.
number of lateralized AVS and number of the patients undergoing adrenalectomy | January 1st 2005 - November 1st 2010
  The number of lateralized AVS will be calculated using different cutoff values for the lateralization index.

CONTACTS AND LOCATIONS:
Overall Officials: GianPaolo Rossi, MD, FACC, Study Director — Dept Clinical and Experimental Medicine (DMCS), University Hospital of Padova, Italy
Locations (20):
- United States (3):
  - Hospital of The University of Pennsylvania, Philadelphia, Philadelphia, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - Medical College of Wisconsin, Menomonee Falls, Wisconsin
- Endocrine Hypertension Research Centre, University of Queensland School of Medicine, Greenslopes Hospital, Brisbane, Australia
- Canada (2):
  - Foothills Medical Centre, University of Calgary, Calgary, Alberta
  - Centre Hospitalier de l'Université de Montreal (CHUM), Montreal, Quebec
- General Faculty Hospital, Prague, Prague, Czechia
- University of Paris, Hopital Européen Georges Pompidou, Paris, France
- Germany (4):
  - Christian J Strasburger, Berlin
  - Heinrich Heine Universität Düsseldorf, Düsseldorf
  - Medizinische Klinik Innenstadt, Munich
  - University Hospital Wuerzburg, Würzburg
- Italy (2):
  - Dept Clinical and Experimental Medicine (DMCS), University Hospital of Padova, Italy, Padua
  - Medicina 2, Dipartimento di Medicina Interna e Specialità Mediche, Azienda Ospedaliera Santa Maria Nuova, Reggio Emilia
- Japan (4):
  - National Hospital Organizatio, Kyoto Medical Center, Kyoto
  - Tohoku University Hospital, Sendai
  - Institute of Clinical Endocrinology, Tokyo Women's Medical University, Tokyo
  - Yokohama Rosai Hospital, Yokohama
- Radboud University Nijmegen Medical Center, Nijmegen, Netherlands
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Funder J, Carey R, Fardella C, Gomez-Sanchez C, Mantero F, Stowasser M, Young W, Montori VM. Withdrawn: Case detection, diagnosis, and treatment of patients with primary aldosteronism: an Endocrine Society clinical practice guideline. Eur J Endocrinol. 2009 Sep 30. doi: 10.1530/EJE-09-0870. Online ahead of print. PMID 19793760
- [Background] Stewart PM, Allolio B. Adrenal vein sampling for Primary Aldosteronism: time for a reality check. Clin Endocrinol (Oxf). 2010 Feb;72(2):146-8. doi: 10.1111/j.1365-2265.2009.03714.x. Epub 2009 Sep 21. No abstract available. PMID 19769616
- [Background] Seccia TM, Miotto D, De Toni R, Pitter G, Mantero F, Pessina AC, Rossi GP. Adrenocorticotropic hormone stimulation during adrenal vein sampling for identifying surgically curable subtypes of primary aldosteronism: comparison of 3 different protocols. Hypertension. 2009 May;53(5):761-6. doi: 10.1161/HYPERTENSIONAHA.108.128553. Epub 2009 Apr 6. PMID 19349554
- [Background] Rossi GP, Pitter G, Bernante P, Motta R, Feltrin G, Miotto D. Adrenal vein sampling for primary aldosteronism: the assessment of selectivity and lateralization of aldosterone excess baseline and after adrenocorticotropic hormone (ACTH) stimulation. J Hypertens. 2008 May;26(5):989-97. doi: 10.1097/HJH.0b013e3282f9e66a. PMID 18398342
- [Background] Mulatero P, Bertello C, Sukor N, Gordon R, Rossato D, Daunt N, Leggett D, Mengozzi G, Veglio F, Stowasser M. Impact of different diagnostic criteria during adrenal vein sampling on reproducibility of subtype diagnosis in patients with primary aldosteronism. Hypertension. 2010 Mar;55(3):667-73. doi: 10.1161/HYPERTENSIONAHA.109.146613. Epub 2010 Feb 1. PMID 20124107
- [Background] Auchus RJ, Wians FH Jr, Anderson ME, Dolmatch BL, Trimmer CK, Josephs SC, Chan D, Toomay S, Nwariaku FE. What we still do not know about adrenal vein sampling for primary aldosteronism. Horm Metab Res. 2010 Jun;42(6):411-5. doi: 10.1055/s-0030-1252060. Epub 2010 Apr 21. PMID 20411476
- [Background] Nishikawa T, Saito J, Omura M. Adrenal venous sampling is absolutely requisite for definitively diagnosing primary aldosteronism as well as for detecting laterality of the adrenal lesion. Hypertens Res. 2007 Nov;30(11):1009-10. doi: 10.1291/hypres.30.1009. No abstract available. PMID 18250546
- [Derived] Pintus G, Seccia TM, Amar L, Azizi M, Riester A, Reincke M, Widimsky J, Naruse M, Kocjan T, Negro A, Kline G, Tanabe A, Satoh F, Rump LC, Vonend O, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Lee BC, Chang CC, Wu VC, Kratka Z, Battistel M, Bagordo D, Caroccia B, Ceolotto G, Rossitto G, Rossi GP. Subtype Identification of Surgically Curable Primary Aldosteronism During Treatment With Mineralocorticoid Receptor Blockade. Hypertension. 2024 Jun;81(6):1391-1399. doi: 10.1161/HYPERTENSIONAHA.124.22721. Epub 2024 Mar 25. PMID 38525605
- [Derived] Rossi GP, Bagordo D, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J, Naruse M, Deinum J, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Rump LC, Vonend O, Willenberg HS, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Lee BC, Chang CC, Wu VC, Kratka Z, Battistel M, Rossitto G, Seccia TM. Unilaterally Selective Adrenal Vein Sampling for Identification of Surgically Curable Primary Aldosteronism. Hypertension. 2023 Oct;80(10):2003-2013. doi: 10.1161/HYPERTENSIONAHA.123.21247. Epub 2023 Jun 15. PMID 37317838
- [Derived] Rossi GP, Crimi F, Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J, Naruse M, Deinum J, Kool LS, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Rump LC, Vonend O, Willenberg HS, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Wu VC, Kratka Z, Barbiero G, Battistel M, Seccia TM. Feasibility of Imaging-Guided Adrenalectomy in Young Patients With Primary Aldosteronism. Hypertension. 2022 Jan;79(1):187-195. doi: 10.1161/HYPERTENSIONAHA.121.18284. Epub 2021 Nov 17. PMID 34878892
- [Derived] Rossi GP, Crimi F, Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J, Naruse M, Deinum J, Schultze Kool L, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Christian Rump L, Vonend O, Willenberg HS, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Cent Wu V, Kratka Z, Barbiero G, Seccia TM, Battistel M. Identification of Surgically Curable Primary Aldosteronism by Imaging in a Large, Multiethnic International Study. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4340-e4349. doi: 10.1210/clinem/dgab482. PMID 34212188
- [Derived] Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J, Naruse M, Deinum J, Schultzekool L, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Rump LC, Vonend O, Willenberg HS, Fuller P, Yang J, Nian Chee NY, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Chang CC, Wu VC, Somloova Z, Maiolino G, Barbiero G, Battistel M, Lenzini L, Quaia E, Pessina AC, Rossi GP. Subtyping of Primary Aldosteronism in the AVIS-2 Study: Assessment of Selectivity and Lateralization. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgz017. doi: 10.1210/clinem/dgz017. PMID 31536622
- [Derived] Rossi GP, Rossitto G, Amar L, Azizi M, Riester A, Reincke M, Degenhart C, Widimsky J Jr, Naruse M, Deinum J, Schultze Kool L, Kocjan T, Negro A, Rossi E, Kline G, Tanabe A, Satoh F, Christian Rump L, Vonend O, Willenberg HS, Fuller PJ, Yang J, Chee NYN, Magill SB, Shafigullina Z, Quinkler M, Oliveras A, Dun Wu K, Wu VC, Kratka Z, Barbiero G, Battistel M, Chang CC, Vanderriele PE, Pessina AC. Clinical Outcomes of 1625 Patients With Primary Aldosteronism Subtyped With Adrenal Vein Sampling. Hypertension. 2019 Oct;74(4):800-808. doi: 10.1161/HYPERTENSIONAHA.119.13463. Epub 2019 Sep 3. PMID 31476901
- [Derived] Rossi GP, Barisa M, Allolio B, Auchus RJ, Amar L, Cohen D, Degenhart C, Deinum J, Fischer E, Gordon R, Kickuth R, Kline G, Lacroix A, Magill S, Miotto D, Naruse M, Nishikawa T, Omura M, Pimenta E, Plouin PF, Quinkler M, Reincke M, Rossi E, Rump LC, Satoh F, Schultze Kool L, Seccia TM, Stowasser M, Tanabe A, Trerotola S, Vonend O, Widimsky J Jr, Wu KD, Wu VC, Pessina AC. The Adrenal Vein Sampling International Study (AVIS) for identifying the major subtypes of primary aldosteronism. J Clin Endocrinol Metab. 2012 May;97(5):1606-14. doi: 10.1210/jc.2011-2830. Epub 2012 Mar 7. PMID 22399502